CLINICAL TRIAL: NCT05717257
Title: Safety and Efficacy of Dapagliflozin in Adult Patients With a Systemic Right Ventricle
Brief Title: Dapagliflozin in Systemic Right Ventricle (DAPA-SERVE)
Acronym: DAPA-SERVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monaldi Hospital (Other)
Responsible Party: Principal Investigator, Flavia Fusco, Medical Doctor, Monaldi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Dapagliflozin Adverse Reaction; Efficacy; Systemic Right Ventricle
Keywords: heart failure; dapagliflozin; systemic right ventricle
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the treatment or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin will be added on top of the standard optimized medical therapy for heart failure and reduced ejection fraction
  Interventions: Drug: Dapagliflozin 10mg Tab
- Control (No Intervention): Participants assigned to this group will continue the standard optimized medical therapy

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10 mg will be added on top of the standard optimized medical therapy for heart failure and reduced ejection fraction
  Arms: Dapagliflozin

SUMMARY:
The purpose of this study is to describe safety and efficacy of Dapaglifozin in adults patients with a systemic right ventricle (congenitally corrected transposition of the great arteries or transposition of the great arteries following arterial switch procedure) and impaired systolic function of the systemic right ventricle.

DETAILED DESCRIPTION:
This is a prospective double arm study aiming to describe safety and efficacy of Dapaglifozin in adults patients with a systemic right ventricle (congenitally corrected transposition of the great arteries or transposition of the great arteries following arterial switch procedure) and impaired systolic function of the systemic right ventricle.

Dapagliflozin will be prescribed in a group of randomly selected patients in addition to the optimized medical therapy for heart failure with reduced ejection fraction.

Changes in quality of life indicators, symptoms, biohumoral markers, exercise capacity and echocardiographic parameters of systolic right ventricular function will be evaluated in comparison with the control group, which will continue standard heart failure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18years
* Optimal medical therapy or at least 3months
* Systemic right ventricle ejection fraction≤40%, assessed on echocardiography

Exclusion Criteria:

* Univentricular physiology
* Systolic blood pressure<90mmHg
* Glomerular filtration rate(GFR)<30ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 1 year
  Absence of any suspected or confirmed adverse events or necessity of drug discontinuation
Nt-proBNP | 1 year
Systemic right ventricle fractional area change | 1 year
Systemic right ventricle global longitudinal strain | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Adult Congenital Heart Disease, Monaldi Hospital, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided